CLINICAL TRIAL: NCT00404534
Title: Dyspeptic Symptoms Evolution After Eradication of Helicobacter Pylori in Patients With Different Endoscopic Findings: a Randomized Double-blind Placebo-controlled Clinical Trial With 12 Months of Follow-up
Brief Title: Helicobacter Eradication Relief of Dyspeptic Symptoms
Acronym: HEROES-12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Aché Laboratórios Farmacêuticos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-422
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2010-03

CONDITIONS: Functional Dyspepsia
Keywords: functional dyspepsia; Helicobacter pylori; Anti-Inflammatory Agents, Non-Steroidal; Gastritis
MeSH Terms: conditions — Gastritis | interventions — Amoxicillin; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Amoxicillin 1000 mg BID, clarythromycin 500 mg BID and Omeprazole 20 mg BID for ten days
  Interventions: Drug: Amoxicillin, Clarythromycin, Omeprazole for ten days
- 2 (Placebo Comparator): Placebo of Amoxicillin 1000 mg BID, placebo of clarythromycin 500 mg BID and Omeprazole 20 mg BID for ten days
  Interventions: Drug: Amoxicillin, Clarythromycin, Omeprazole for ten days

INTERVENTIONS:
Drug: Amoxicillin, Clarythromycin, Omeprazole for ten days — Amoxicillin 1000 mg BID, clarythromycin 500 mg BID for ten days in the experimental group and placebo of Amoxicillin 1000 mg BID and placebo of clarythromycin 500 mg BID in the placebo comparator. Both groups receive omeprazole 20 mg bid for 10 days.

SUMMARY:
A double-blind clinical trial investigating if a sub-group of functional dyspeptic patients without any use of NSAID or gastric erosions could have a better evolution of their dyspeptic symptoms after Helicobacter eradication than the placebo control group

DETAILED DESCRIPTION:
Objective: investigate if a sub-group of functional dyspeptic patients without any use of NSAID or gastric erosions could have a better evolution of their dyspeptic symptoms after Helicobacter eradication than the placebo control group

Design: A randomized double-blind placebo controlled clinical trial

Inclusion Criteria: Patients with more than 18 years, Functional dyspepsia accordingly Rome III criteria, Helicobacter pylori infection by two diagnostic tests

Exclusion Criteria: No concordance with informed consent; Pregnant woman or breast feeding or no trust anticonceptional method; Structural gastrointestinal abnormalities except gastritis, duodenitis or hiatal hernia; Previous treatment for Helicobacter pylori infection; Previous surgery on esophagus, stomach or duodenum; Hypersensitivity to the drugs in study; Proton pump inhibitor use in the previous 15 days; H2-antagonists use in the previous 07 days; Antibiotics use in the previous 30 days; Patients unable to answer the study questionnaires; Alcohol abuse; Drug use; Serious comorbidities; Biliary colic; Irritable bowel syndrome; Gastroesophageal Reflux Disease

Interventions: amoxicillin, clarythromycin, omeprazole for 10 days

Control: Placebo

Outcomes:

Primary: Proportion of patients with 50% reduction of baseline symptoms score measured by the validated Porto Alegre Dyspeptic Symptoms Questionnaire Secondary: Proportion of patients with 100% reduction of baseline symptoms score measured by the validated Porto Alegre Dyspeptic Symptoms Questionnaire; Need of rescue medication; Median difference of score between groups; Mean SF-36 scores evolution between groups; Lost of productivity measured by WPAI between groups

Visits: screening, baseline, 4, 8, 12 months

Endoscopic evaluation: screening, 12 months

Helicobacter detection methods: urease, histology (3 pathologists) performed at screening and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 18 years
* Functional dyspepsia accordingly Rome III criteria
* Helicobacter pylori infection by two diagnostic tests

Exclusion Criteria:

* No concordance with informed consent
* Pregnant woman or breast feeding or no trust anticonceptional method
* Structural gastrointestinal abnormalities except gastritis, duodenitis or hiatal hernia
* Previous treatment for Helicobacter pylori infection
* Previous surgery on esophagus, stomach or duodenum
* Hypersensitivity to the drugs in study
* Proton pump inhibitor use in the previous 15 days
* H2-antagonists use in the previous 07 days
* Antibiotics use in the previous 30 days
* Patients unable to answer the study questionnaires
* Alcohol abuse
* Drug use
* Serious comorbidities
* Biliary colic
* Irritable bowel syndrome
* Gastroesophageal Reflux Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with 50% reduction of baseline symptoms score measured by the validated Porto Alegre Dyspeptic Symptoms Questionnaire | the last visit among the antecipated visits (4, 8 and 12 months)

SECONDARY OUTCOMES:
Proportion of patients with 100% reduction of baseline symptoms score measured by the validated Porto Alegre Dyspeptic Symptoms Questionnaire | the last visit among the antecipated visits (4, 8 and 12 months)
Need of rescue medication | 4, 8 and 12 months
Median difference of score between groups | the last visit among the antecipated visits (4, 8 and 12 months)
Mean SF-36 scores evolution between groups | 12 months
Lost of productivity measured by WPAI between groups | 12 months
Adverse Events | 4 , 8 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Luiz E Mazzoleni, MD, MsC, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre, Universidade Federal do Rio Grande do Sul; Carlos F Francesconi, MD, PhD, Study Chair — Hospital de Clinicas de Porto Alegre, Universidade Federal do Rio Grande do Sul; Guilherme B Sander, MD, MsC, Study Chair — Hospital de Clinicas de Porto Alegre, Universidade Federal do Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Mazzoleni LE, Sander GB, Ott EA, Barros SG, Francesconi CF, Polanczyk CA, Wortmann AC, Theil AL, Fritscher LG, Rivero LF, Cartell A, Edelweiss MI, Uchoa DM, Prolla JC. Clinical outcomes of eradication of Helicobacter pylori in nonulcer dyspepsia in a population with a high prevalence of infection: results of a 12-month randomized, double blind, placebo-controlled study. Dig Dis Sci. 2006 Jan;51(1):89-98. doi: 10.1007/s10620-006-3090-6. PMID 16416218
- [Background] Ott EA, Mazzoleni LE, Edelweiss MI, Sander GB, Wortmann AC, Theil AL, Somm G, Cartell A, Rivero LF, Uchoa DM, Francesconi CF, Prolla JC. Helicobacter pylori eradication does not cause reflux oesophagitis in functional dyspeptic patients: a randomized, investigator-blinded, placebo-controlled trial. Aliment Pharmacol Ther. 2005 May 15;21(10):1231-9. doi: 10.1111/j.1365-2036.2005.02461.x. PMID 15882244
- [Background] Sander GB, Mazzoleni LE, Francesconi CF, Wortmann AC, Ott EA, Theil A, Da Cruz PV, Da Silva AC, Oliveira L, Beheregaray S, Matioti S, Somm G, Goldim JR. Development and validation of a cross-cultural questionnaire to evaluate nonulcer dyspepsia: the Porto Alegre Dyspeptic Symptoms Questionnaire (PADYQ). Dig Dis Sci. 2004 Nov-Dec;49(11-12):1822-9. doi: 10.1007/s10620-004-9578-z. PMID 15628711
- [Derived] Mazzoleni LE, Sander GB, Francesconi CF, Mazzoleni F, Uchoa DM, De Bona LR, Milbradt TC, Von Reisswitz PS, Berwanger O, Bressel M, Edelweiss MI, Marini SS, Molina CG, Folador L, Lunkes RP, Heck R, Birkhan OA, Spindler BM, Katz N, Colombo Bda S, Guerrieri PP, Renck LB, Grando E, Hocevar de Moura B, Dahmer FD, Rauber J, Prolla JC. Helicobacter pylori eradication in functional dyspepsia: HEROES trial. Arch Intern Med. 2011 Nov 28;171(21):1929-36. doi: 10.1001/archinternmed.2011.533. PMID 22123802
- [Derived] Sander GB, Mazzoleni LE, Francesconi CF, Balbinotto G, Mazzoleni F, Wortmann AC, Cardoso Ide Q, Klamt AL, Milbradt TC; Helicobacter Eradication Relief of Dyspetic Symptoms Trial Investigators. Influence of organic and functional dyspepsia on work productivity: the HEROES-DIP study. Value Health. 2011 Jul-Aug;14(5 Suppl 1):S126-9. doi: 10.1016/j.jval.2011.05.021. PMID 21839884
- See also: Official Homepage of Site that is Conducting the Study — http://www.hcpa.ufrgs.br